CLINICAL TRIAL: NCT02972918
Title: Preoperative Optimization Levosimendan in Heart Failure Patients Undergoing Hip Fracture
Brief Title: Preoperative levosimendán and Hip Fracture
Acronym: OPL
Status: Completed | Type: Observational
Sponsor: Hospital Universitario de Canarias (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, María del Carmen Martín Lorenzo, Dr, Hospital Universitario de Canarias
Other Study IDs: MML-LEV-2013-01
Record Dates: First submitted 2016-11-14; First posted 2016-11-25 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Ventricular Dysfunction, Left; Hip Fracture
MeSH Terms: conditions — Ventricular Dysfunction, Left; Hip Fractures | interventions — Simendan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Levosimendan: At least 12 hours before surgery: Infusion of levosimendan (0,1 mcg/kg/min). 24 hours of infusion without a bolus.
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — 24h preoperative infusion of levosimendan (0,1 mcg/Kg/min)
  Other Names: Simdax.

SUMMARY:
The purpose of this study is to evaluate whether preoperative optimization with levosimendan in heart failure patients undergoing hip fracture surgery improves haemodynamic and tissue perfusion parameters.

DETAILED DESCRIPTION:
Hip fracture is a very predominant entity in elderly patients and it is one of the most frequent cause of admission in a hospital.

Elderly patients undergoing surgery for hip fracture have a high risk of morbidity and mortality in the postoperative. Several studies have shown that there is a high risk of cardiovascular complications in this group of patients and 3-months mortality is 15-20%. One of the causes of this high morbidity and mortality is the high incidence of chronic cardiac failure in this patients. The goal of the present study is to evaluate if the optimization of preoperative cardiac function with levosimendan in patients with left ventricular ejection fraction < 45% can improve haemodynamic and the tissue perfusion values, and reduce cardiac morbidity and mortality 3 months postoperatively.

Following written consent, the patients with left ventricular ejection fraction < 45% will be admitted in the resuscitation and anaesthesia room where they will receive a levosimendan intravenous injection undergoing a strict haemodynamic vigilance.

Before the levosimendan intravenous injection the patients firs have an echocardiography to evaluate myocardial function, NT-proBNP. Subsequently, an arterial line is inserted and optimization achieved by using this arterial line connected to a ProAQT sensor system ( PULSION , Edwards). The system uses pulse wave analysis to assess several parameters including: stroke volume index (SVI), cardiac index (CI), systemic vascular resistance index (SVRI), cardiac power index (CPI).The levosimendan will be administered like a continues injection during 24 hours (0,1 mcg/kg/min) without initial dose. Following the optimization the patients will be transferred to the operating room in the next 3 days and will come back to the resuscitation and anaesthesia room where they will stay 24 hours more if there is no any complication.

All the cardiac complications will be documented and follw-up will be done by after 30 days and 3 months postoperative.

The patients will be selected for more than 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients due to undergo urgent of hip fracture.
2. Patients with cardiac failure (EF < 45 %).
3. Decompensated heart failure.
4. Informed consent provided by the patient.

Exclusion Criteria:

1. <18 years old
2. Emergency surgery
3. Serious aortic stenosis (< 1 cm2)
4. Sustained ventricular tachycardia or atrial fibrillation >140
5. Earlier episodes of "torsades depointes"
6. Systolic blood pressure < 85 mmHg
7. Serious kidney failure (GFR < 30 ml/min)
8. Serious liver failure (known class C Child-Pugh score)
9. Allergy levosimendan

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with chronic heart failure of any etiology with hip fracture that present an acute descompendation of their chronic heart failure and need inotropes because of the conventional treatment is not enough
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The effects of Levosimendan on left ventricular function. | Baseline and every 24 hours postoperative, 48 h postoperative, and 7 days and after 30 days postoperative.
  Changes of left ventricular function as assessed transthoracic.
Change in cardiac index | 48 hours after start of iv infusion
  Measured through arterial pulse wave analysis. A baseline measurement is done before infusion is started

SECONDARY OUTCOMES:
Changes in transport and tissue perfusion of oxygen | 1 to 2 day postoperative
  measured by arterial and venous blood gases
Changes in renal function | 1 to 7 days postoperative
  Proportion of subjects who develop AKIN stage 1 (increase > 0.3 mg/dl or > 25% in serum creatinine from previous visit)
Changes in NT-proBNP and troponin I | 24 hours postoperative, 48 h postoperative, 72 h postoperative, and 168 h postoperative
  Plasma NT-proBNP levels were measured
Number of patients with adverse. | 30 days postoperative
  Development of arrhythmias
Number of patients with adverse. | 30 days postoperative
  Occurence of nausea/vomiting
Number of patients with adverse event. | 30 days postoperative
  Occurence of headache
Use of high inotropes (dopamine, Norepinephrine) | after 12 hours, after 48 hours and every 24 hours if still in the PO-Unit
  during postoperative unit stay.
morbidity | 3 months
  All cause
Major adverse cardiovascular events | 1st-30th postoperative day
  Perioperative heart failure infarction, stroke
Time on mechanical ventilation | 1st-30th postoperative day
  Perioperative heart failure infarction, stroke
mortality | measured at 3 months
  All cause
Perioperative mortality | 7 days postoperative
  All cause

CONTACTS AND LOCATIONS:
Overall Officials: María del Carmen Martín Lorenzo, MD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna, S/C Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cauley JA, Thompson DE, Ensrud KC, Scott JC, Black D. Risk of mortality following clinical fractures. Osteoporos Int. 2000;11(7):556-61. doi: 10.1007/s001980070075. PMID 11069188
- [Result] Center JR, Nguyen TV, Schneider D, Sambrook PN, Eisman JA. Mortality after all major types of osteoporotic fracture in men and women: an observational study. Lancet. 1999 Mar 13;353(9156):878-82. doi: 10.1016/S0140-6736(98)09075-8. PMID 10093980
- [Result] Pedersen SJ, Borgbjerg FM, Schousboe B, Pedersen BD, Jorgensen HL, Duus BR, Lauritzen JB; Hip Fracture Group of Bispebjerg Hospital. A comprehensive hip fracture program reduces complication rates and mortality. J Am Geriatr Soc. 2008 Oct;56(10):1831-8. doi: 10.1111/j.1532-5415.2008.01945.x. PMID 19054201
- [Result] Ponschab M, Hochmair N, Ghazwinian N, Mueller T, Plochl W. Levosimendan infusion improves haemodynamics in elderly heart failure patients undergoing urgent hip fracture repair. Eur J Anaesthesiol. 2008 Aug;25(8):627-33. doi: 10.1017/S0265021508004080. Epub 2008 Apr 11. PMID 18405408